CLINICAL TRIAL: NCT00920270
Title: Efficacy and Safety of Nebulized Colistin for Adjunctive Therapy of Hospital-Acquired Pneumonia Caused by Gram Negative Bacteria
Brief Title: Nebulized Colistin for Hospital-Acquired Pneumonia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mahidol University (Other)
Responsible Party: Visanu Thamlikitkul, Siriraj Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Siriraj CEU 50-002
Record Dates: First submitted 2009-06-11; First posted 2009-06-15 (Estimated); Last update posted 2009-06-15 (Estimated); Status verified 2006-06

CONDITIONS: Pneumonia
Keywords: Hospital-Acquired Pneumonia; Gram Negative Bacteria
MeSH Terms: conditions — Pneumonia; Healthcare-Associated Pneumonia | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- antibiotic (Active Comparator): conventional antibiotics
  Interventions: Drug: antibiotics
- colistin group (Experimental): nebulized colistin
  Interventions: Drug: nebulized colistin

INTERVENTIONS:
Drug: nebulized colistin — nebulized colistin 75 mg every 12 hours
  Arms: colistin group
Drug: antibiotics — conventional parenteral antibiotics
  Arms: antibiotic

SUMMARY:
Nebulized Colistin for Adjunctive Therapy of Hospital-Acquired Pneumonia caused by Gram Negative Bacteria should be more effective than conventional therapy

DETAILED DESCRIPTION:
Randomized Controlled Clinical Trial in hospitalized adult patients with hospital-acquired pneumonia. The patients are allocated to conventional group or nebulized colistin group. The conventional group receives conventional antibiotics whereas the nebulized colistin group receives nebulized colistin in addition to conventional antibiotics. The outcomes are clinical response and microbiological responses.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age>18 years) hospitalized patient with hospital-acquired pneumonia due to Gram negative bacteria

Exclusion Criteria:

* pregnancy
* lactating woman
* colistin allergy
* severe renal impairment
* epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2006-06; Primary Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Clinical response | 14 days after Treatment

SECONDARY OUTCOMES:
Microbiological response and safety | 14 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Visanu Thamlikitkul, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkok, Bangkok, Thailand